CLINICAL TRIAL: NCT05789329
Title: Non-Inferiority Trial of Trauma Informed Guilt Reduction Therapy (TrIGR) for PTSD
Brief Title: Non-Inferiority Trial of TrIGR for PTSD
Acronym: TrIGR/CPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBP-003-22S; I01CX002584 (NIH)
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: PTSD
Keywords: PTSD; trauma; moral injury; intervention; guilt; shame
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to Trauma Informed Guilt Reduction Therapy (TrIGR) or Cognitive Processing Therapy (CPT).
Who Masked: Outcomes Assessor
Masking Description: A computer-generated masked randomization sequence will be provided and held by a statistician not otherwise involved in the study. Randomization will be stratified by site and gender.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trauma Informed Guilt Reduction Therapy (TrIGR) (Experimental): behavioral intervention aimed to reduce trauma-related guilt and shame
  Interventions: Behavioral: Trauma Informed Guilt Reduction Therapy
- Cognitive Processing Therapy (CPT) (Active Comparator): behavioral intervention aimed at reducing PTSD symptoms
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Trauma Informed Guilt Reduction Therapy — behavioral intervention aimed to reduce trauma-related guilt and shame
  Other Names: TrIGR
  Arms: Trauma Informed Guilt Reduction Therapy (TrIGR)
Behavioral: Cognitive Processing Therapy — behavioral intervention aimed at reducing PTSD symptoms
  Other Names: CPT
  Arms: Cognitive Processing Therapy (CPT)

SUMMARY:
Trauma-related guilt is common and impairing among trauma survivors, particularly among Veterans with posttraumatic stress disorder (PTSD). The investigators' work shows that a brief treatment targeting trauma-related guilt, Trauma Informed Guilt Reduction Therapy (TrIGR), can reduce guilt and PTSD and depression symptoms. Whether TrIGR is no less effective than longer, more resource heavy PTSD treatments disseminated by by VA, like cognitive processing therapy (CPT), is the next critical question that this study will seek to answer. 158 Veterans across two VA sites will be randomized to TrIGR or CPT to evaluate changes in PTSD, depression, guilt and shame symptoms across the two treatments.

DETAILED DESCRIPTION:
Trauma-related guilt is common and impairing among trauma survivors, particularly among treatment seeking Veterans with posttraumatic stress disorder (PTSD). Although evidence-based trauma-focused PTSD treatments such as Cognitive Processing Therapy (CPT) are effective to treat PTSD and trauma-related guilt, many still experience symptoms or maintain their diagnosis after treatment, and dropout from these generally 12+ session protocols is high. Veterans show lower response and higher dropout than others with PTSD. Delivering protocols that are generally 12 or more sessions challenges the Veterans Affairs (VA) healthcare system given high demand for mental health care. For these reasons, additional and less burdensome approaches are needed. Brief treatment that targets mechanisms that are distressing and associated with multiple problems and disorders may be an understudied but promising way to treat PTSD and other posttraumatic psychopathology. The investigators' work shows that a brief treatment targeting trauma-related guilt and shame, Trauma Informed Guilt Reduction Therapy (TrIGR), can reduce guilt, PTSD, depression, and distress among Veterans and help them reengage with activities they find meaningful. Whether TrIGR is no less effective than longer, more resource heavy evidence-based PTSD treatments disseminated across by VA, like CPT, is the next critical question.

The proposed randomized clinical trial (RCT) will be the first non-inferiority trial of TrIGR and the first to compare TrIGR to a first tier PTSD treatment, specifically CPT. It will also be the first to evaluate TrIGR with Veterans from all eras with guilt from any type of traumas, as the investigators previous work was exclusively with Veterans of the conflicts in Iraq and Afghanistan with deployment-related traumas. 158 Veterans across two VA sites will be randomized to TrIGR or CPT. Exclusion criteria will be minimal so that generalizability will be high. Treatment will be delivered in VA mental health clinics. The primary aim is to evaluate if TrIGR is non-inferior to CPT in reducing PTSD symptom severity among Veterans with PTSD who endorse trauma-related guilt. Secondary aims are to evaluate TrIGR's non-inferiority relative to CPT regarding depression severity. The investigators will explore potential mechanisms of treatment, such as the relationship between change in guilt and shame change in PTSD symptoms. The study is critical to establish whether TrIGR is effective for a much larger group of Veterans and whether it is as effective as longer treatments already available in VA to inform if TrIGR warrants further study and dissemination in VA.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veterans age 18 or older;
* meets diagnostic criteria for PTSD or subthreshold PTSD;
* a score of 2 or higher ("true" to "extremely true") on feeling trauma-related guilt much or all of the time or scoring 3 or higher ("very true" or "extremely true") on at least one guilt cognition factor (hindsight bias/responsibility, wrongdoing, or lack of justification) on the Trauma Related Guilt Inventor.
* not currently receiving trauma-focused treatment such as CPT or PE; and
* willingness to attend psychotherapy and assessment sessions.

Exclusion Criteria:

* Impaired mental status as measured by the Montreal Cognitive Assessment (MoCA) (score < 21) and confirmed by a neuropsychologist,
* Veterans with significant current risk of suicidal/homicidal behavior will be referred to more appropriate treatment;
* Current severe substance use disorder (in the past two months) based on DSM-5 criteria;
* Current unmanaged psychosis or mania;
* life threatening or unstable medical illness; or
* inability to read.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
change in Clinician Administered PTSD Scale - 5 (CAPS-5) | baseline to 28 weeks later
  Clinician Administered PTSD Scale - 5 (CAPS-5) - score range 0 - 80; higher scores are indicative of more severe PTSD symptoms. Reduction in scores is considered a positive outcome.

SECONDARY OUTCOMES:
change in Patient Health Questionnaire - 9 (PHQ-9) | baseline to 28 weeks later
  change in Patient Health Questionnaire - 9 (PHQ-9) - score ranges 0-27. higher scores are indicative of more severe depressive symptoms. Reduction in scores is considered a positive outcome.
Trauma Related Guilt Inventory (TRGI) | baseline to 28 weeks later
  Trauma Related Guilt Inventory (TRGI) - score ranges 0-4. higher scores are indicative of more severe trauma-related guilt. Reduction in scores is considered a positive outcome.
Trauma Related Shame Inventory (TRSI) | baseline to 28 weeks later
  Trauma Related Shame Inventory (S) - score ranges 0-72. higher scores are indicative of more severe trauma-related shame. Reduction in scores is considered a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sonya B. Norman, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset without personal identifiers will be generated and shared with those who request and are granted access (see access criteria). Any HIPAA identifiers, or combinations of variables that could be used for re-identification, will be excluded, as will any proprietary information. The plan does not include any access to individually identifiable or proprietary data. Therefore, this plan will ensure the protection of personal privacy, the confidentiality of individually identifiable private information, and the security of proprietary data and information.
Supporting Information: Study Protocol
Time Frame: After publication of the primary outcome paper.
Access Criteria: Requests for access must be made in writing signed by a requester from the United States and include an email address for delivery and an assurance that the recipient will not attempt to identify or re-identify any individual. The request should reference the publication underlying the request.